CLINICAL TRIAL: NCT03262597
Title: Beverage Hydration Index of Three Commercial Oral Rehydration Therapy ORT Beverages
Brief Title: "Beverage Hydration Index" of Commercial Therapeutic Beverages
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sonoma State University (Other)
Collaborators: Entrinsic Bioscience Inc. (Industry)
Responsible Party: Principal Investigator, Kurt Sollanek, Assistant Professor, Sonoma State University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: IRB Application #2667
Record Dates: First submitted 2017-08-23; First posted 2017-08-25 (Actual); Last update posted 2018-03-07 (Actual); Status verified 2018-03

CONDITIONS: Healthy
Keywords: fluid balance; dehydration; rehydration; electrolytes; urine
MeSH Terms: conditions — Dehydration | interventions — gatorade; Water

STUDY DESIGN:
Intervention Model Description: Repeated-measures design with generalized latin square arrangement. Each participant will complete 4 separate trials.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Beverage Hydration Index of beverages (Experimental): Subjects will consume 4 different beverages to obtain the beverage hydration index.
  Interventions: Other: enterade; Other: Pedialyte; Other: Gatorade; Other: Water

INTERVENTIONS:
Other: enterade — Subjects will consume enterade, which is an amino acid-based oral rehydration solution.
Other: Pedialyte — Subjects will consume Pedialyte
Other: Gatorade — Subjects will consume Gatorade
Other: Water — Subjects will consume water as the control beverage

SUMMARY:
The "beverage hydration index" (BHI) assesses the hydration potential of any consumable fluid relative to water. The BHI is a relatively new metric. Our purpose was to assess the BHI of beverages never previously tested, including an amino acid-based oral rehydration solution (AA-ORS), a glucose-containing ORS (G-ORS) and a sports drink (SD) compared to water (control).

DETAILED DESCRIPTION:
The "Beverage Hydration Index" (BHI) was created to assess the degree to which beverages "hydrate", by measuring fluid retention after ingesting a 1 liter bolus and comparing it to water. Drinks with carbohydrates and electrolytes would traditionally be expected to score higher on the BHI due to glucose-sodium cotransport at the gut and osmolality approaching isotonicity with blood. One recent study reported that an oral rehydration solution (ORS) scored better than water, but a "sports drink" did not. No "optimal" BHI beverage composition has been described, nor has an optimal osmolality. Recently, a hypotonic amino acid-based rehydration beverage was developed to take advantage of amino acid-sodium cotransport, thus obviating the need for carbohydrate. However, the BHI of this beverage has not yet been assessed. The purpose of this investigation was to assess the hydration potential of this novel beverage in comparison to a commercially available carbohydrate-containing sports drink and oral rehydration solution.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male or female
* Aged 18-35
* BMI 18-27 kg/m2
* No known cardiovascular, renal or metabolic disease
* Moderately active
* Moderate alcohol use

Exclusion Criteria:

* Overweight or obese (BMI >27 kg/m2)

  * Competitive athletes during competition season
  * Current or former cardiovascular, renal or metabolic disease
  * Habitual consumption of alcohol (>21 units/week) or regular (>1/week) high (10 units) intake*
  * History of psychiatric illness
  * Actively seeking to gain or lose weight
  * Currently taking prescribed medication

    * Example, a 750 ml bottle of wine at 12% ABV contains 0.750 Liters * 12 = 9 units

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 46 (Actual)
Dates: Start 2017-02-17 (Actual); Primary Completion 2017-04-14 (Actual); Study Completion 2017-04-14 (Actual)

PRIMARY OUTCOMES:
Beverage hydration index | 4 hours
  beverage hydration index

CONTACTS AND LOCATIONS:
Overall Officials: Kurt J Sollanek, Ph.D., Principal Investigator — Sonoma State University
Locations (1):
- Sonoma State Univrsity, Rohnert Park, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Sollanek KJ, Tsurumoto M, Vidyasagar S, Kenefick RW, Cheuvront SN. Neither body mass nor sex influences beverage hydration index outcomes during randomized trial when comparing 3 commercial beverages. Am J Clin Nutr. 2018 Apr 1;107(4):544-549. doi: 10.1093/ajcn/nqy005. PMID 29635499